CLINICAL TRIAL: NCT01497782
Title: Impact of Instructor Feedback on Performance in a Virtual Reality Simulator: A Randomized, Controlled Trial
Brief Title: The FEEDBACK Trial, a Randomized Controlled Trial
Acronym: Feedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Jeanett Oestergaard, MD, PhD fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-3-2010-082 FEEDBACK
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Laparoscopic Proficiency
Keywords: virtual reality, simulator, feedback, laparoscopy, training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instructor feedback (Experimental): Intervention group who receives up to three sessions of instructor feedback during completion of a predefined proficiency level on a laparoscopic virtual reality simulator.
  Interventions: Other: Instructor feedback
- No instructor feedback (No Intervention): Control group who did not receive instructor feedback during completion of a predefined proficiency level on a laparoscopic virtual reality simulator.

INTERVENTIONS:
Other: Instructor feedback — Intervention group who receives up to three sessions of instructor feedback during completion of a predefined proficiency level on a laparoscopic virtual reality simulator.
  Arms: Instructor feedback

SUMMARY:
With a worldwide proliferation of simulation centers, it is essential to explore the optimal setting for laparoscopic training and investigate different learning approaches, e.g. a self-directed approach. Therefore, the researchers investigated the following in a randomized controlled trial: the impact of instructor feedback vs. an independent, self-directed approach when training a complex operational task on a laparoscopic virtual reality simulator.

The study hypothesis is that instructor feedback has a pivotal effect on surgical skills when training on a virtual reality simulator.

DETAILED DESCRIPTION:
For virtual reality (VR) simulation the benefits are clear; the drawbacks are less clear. Throughout the last decade several studies have found a positive effect on the learning curve as well as improvement of basic psychomotor skills in the operating room after VR training. VR simulators offer standardized and reproducible laparoscopic tasks, ranging from simple basic skills training to full procedures such as a cholecystectomy or salpingectomy. Despite the now well-established advantages of VR simulators, the majority of surgical and gynecological departments encounter hurdles when implementing this form of training in the surgical education. This is mainly due to lack of knowledge concerning the time and human resources/cost needed to train novice surgeons to an adequate level.

This randomized trial investigates whether instructor feedback is pivotal for the trainee when training operational tasks (a laparoscopic salpingectomy) on a VR simulator. The VR simulator used in this trial is the LapSim from Surgical Science, Sweden. Instructor feedback consists of standardized feedback for ten minutes and with a maximum of three optional feedback sessions; the trainees (in the intervention group) decides them selves when they want a feedback session. The trainees in both the control group and the intervention group have to reach a predefined proficiency level on the VR simulator within 8 weeks with 3-hour training sessions each time. Furthermore, the trial focuses on different learning approaches, e.g. a self-directed approach and an independent approach.

The randomization process will take place at a central unit; Copenhagen Trial Unit, Denmark. Stratification variables are: 1)Gender 2)Computer game experience (less that 20 hours annually)

ELIGIBILITY:
Inclusion Criteria:

* Medical student at Copenhagen University with passed bachelor degree
* Signed informed consent

Exclusion Criteria:

* Prior experience with surgical virtual reality simulators
* > 3 independent laparoscopic procedures
* Not fluent in the Danish language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Repetitions | 8 weeks
  Number of repetitions to complete a predefined proficiency level on a laparoscopic virtual reality simulator

SECONDARY OUTCOMES:
Time | 8 weeks
  Time to complete a predefined proficiency level on a laparoscopic virtual reality simulator.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanett Oestergaard, MD, Principal Investigator — Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen Ø, Denmark
Locations (1):
- Rigshospitalet, University Hospital of Copenhagen, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Larsen CR, Soerensen JL, Grantcharov TP, Dalsgaard T, Schouenborg L, Ottosen C, Schroeder TV, Ottesen BS. Effect of virtual reality training on laparoscopic surgery: randomised controlled trial. BMJ. 2009 May 14;338:b1802. doi: 10.1136/bmj.b1802. PMID 19443914
- [Background] Larsen CR, Grantcharov T, Aggarwal R, Tully A, Sorensen JL, Dalsgaard T, Ottesen B. Objective assessment of gynecologic laparoscopic skills using the LapSimGyn virtual reality simulator. Surg Endosc. 2006 Sep;20(9):1460-6. doi: 10.1007/s00464-005-0745-x. Epub 2006 Jul 3. PMID 16823649
- [Derived] Bjerrum F, Maagaard M, Led Sorensen J, Rifbjerg Larsen C, Ringsted C, Winkel P, Ottesen B, Strandbygaard J. Effect of instructor feedback on skills retention after laparoscopic simulator training: follow-up of a randomized trial. J Surg Educ. 2015 Jan-Feb;72(1):53-60. doi: 10.1016/j.jsurg.2014.06.013. Epub 2014 Aug 16. PMID 25139606
- [Derived] Strandbygaard J, Bjerrum F, Maagaard M, Winkel P, Larsen CR, Ringsted C, Gluud C, Grantcharov T, Ottesen B, Sorensen JL. Instructor feedback versus no instructor feedback on performance in a laparoscopic virtual reality simulator: a randomized trial. Ann Surg. 2013 May;257(5):839-44. doi: 10.1097/SLA.0b013e31827eee6e. PMID 23295321
- [Derived] Oestergaard J, Bjerrum F, Maagaard M, Winkel P, Larsen CR, Ringsted C, Gluud C, Grantcharov T, Ottesen B, Soerensen JL. Instructor feedback versus no instructor feedback on performance in a laparoscopic virtual reality simulator: a randomized educational trial. BMC Med Educ. 2012 Feb 28;12:7. doi: 10.1186/1472-6920-12-7. PMID 22373062